CLINICAL TRIAL: NCT03578705
Title: Longitudinal Evaluation of Muscle Quality in Patients With Fractures - A Prospective Observational Study
Brief Title: Muscle Quality and Percentage of Fat Following a Lower Limb Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Edward Harvey, Professor of Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 15-056-MUHC
Record Dates: First submitted 2017-08-02; First posted 2018-07-06 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Lower Limb Injury; Injury Trauma
Keywords: Orthopedic trauma
MeSH Terms: conditions — Leg Injuries; Accidental Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Electrical Impedance Myography unit or "EIM"

SUMMARY:
The aim of the study is to longitudinally evaluate patient muscle quality in trauma patients with bed rest or altered weight-bearing with the help of a consumer approved non-proprietary muscle impedance-measuring device. Secondary objectives are to identify patient characteristics or treatment protocols that are predictive of poor muscle quality.

DETAILED DESCRIPTION:
The study investigators will identify eligible patients through patient consultations from the Emergency Room. There are 100 patients expected to be enrolled in the study. This study will be carried out at the Montreal General Hospital. Inclusion criteria include patients that have had a trauma requiring admission to orthopedic surgery, that have the ability and willingness to participate that were in a steady state medical condition before trauma.

Although the study investigators may discuss the study with the patient, the consent and enrolment will be performed exclusively by the study assistant who is not directly implicated in the patient's care.

This is an observational study, therefore, there will be no randomization and no study intervention.

The following baseline patient characteristics will be recorded for each enrolled participant: age, sex, occupation, smoker, medical comorbidities, AO classification of the fractures and muscle trauma, the date of the injury and date of the surgery if performed.

A consumer approved non-proprietary muscle impedance-measuring device (Electrical Impedance Myography unit or "EIM") will be applied to the muscle groups of interest. The device is self-contained, battery-powered and certified for use on humans. When applied to the skin, a very weak electrical current is passed between the outer two electrodes. This current is high frequency and alternating in nature. As the current moves through the skin, the subcutaneous fat and the muscle, it loses a little bit of energy due to the resistance of the tissue and this change is then measured. This will be done as soon as possible after the trauma and admission during a daytime visit. The EIM will be used every two days until discharge or the patient has reached a recovery plateau in a physical rehabilitation program. Patients' muscle quality will also be measured at each follow-up visit for 100 weeks and patients will be asked to complete two questionnaires.

Each patient will have a unique identification number used to link the patient information, device and data together.

It is expected for most patients to have decreasing muscle quality and increasing fat percentage as a result of deconditioning. There is no longitudinal data on the time period over which this would occur. There is also little data on how recovery occurs after the period of healing.

This study utilizes new technology that permits objective insight into the post-operative period by providing qualitative measurements. It has been used previously in clinical studies on patients with neuromuscular degenerative disease with reproducible and consistent results. The research team anticipates being able to pinpoint specific targets for mobilization goals and rehabilitation techniques depending on the time frame and muscle groups involved with deconditioning.

ELIGIBILITY:
Inclusion Criteria:

* Trauma requiring admission to orthopedic surgery because of a lower limb injury
* Ability and willingness to participate
* Steady state medical condition before trauma

Exclusion Criteria:

* Age <18
* Pre-existing condition that caused pain or limited weight-bearing on either lower extremity before sustaining trauma (for example the use of walking aids)
* Pre-existing medical conditions that will confound the study outcomes (muscle conditions) and are known to prevent return to function
* Pregnancy
* Implanted electrical device such as heart pacemakers

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any adult patient admitted at the Montreal General Hospital for orthopedic surgery because of a lower limb injury preventing them to walk without aid for a certain time.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Quality | Every two-day while in bed rest at the hospital and at every follow-up visit up to 100 weeks after injury
  The muscle quality number given by the device is a number given by the company making the device with an arbitrary standard.
Percentage of Fat Measurement | Every two-day while in bed rest at the hospital and at every follow-up visit up to 100 weeks after injury
  The percentage of fat is given by the device

CONTACTS AND LOCATIONS:
Overall Officials: Edward Harvey, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
We will share the results from the collected data in a publication. However, we will not share individual participant data for reasons of confidentiality.